CLINICAL TRIAL: NCT00041925
Title: A Phase III, Multi-Center Randomized, Double-Blind, Placebo-Controlled Trial of the Ex Vivo Treatment With CGT003 of Peripheral Vein Grafts in Patients Undergoing Peripheral Arterial Bypass Graft Procedures
Brief Title: Prevention of Autogenous Vein Graft Failure in Peripheral Artery Bypass Procedures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anesiva, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CGT003-03
Record Dates: First submitted 2002-07-18; First posted 2002-07-22 (Estimated); Last update posted 2005-07-15 (Estimated); Status verified 2005-07

CONDITIONS: Peripheral Vascular Diseases; Arterial Occlusive Diseases; Ischemia; Graft Occlusion, Vascular; Hyperplasia
Keywords: atherosclerotic vascular disease; chronic critical limb ischemia; neointimal hyperplasia; peripheral vein bypass; infra-inguinal bypass grafting surgery; graft stenosis; occluded grafts
MeSH Terms: conditions — Peripheral Vascular Diseases; Arterial Occlusive Diseases; Ischemia; Graft Occlusion, Vascular; Hyperplasia; Atherosclerosis

INTERVENTIONS:
Drug: CGT003 (E2F Duplex Decoy)

SUMMARY:
The purpose of this study is to determine the efficacy of graft pretreatment with the E2F decoy, CGT003, as compared to placebo, on the occurrence of graft failure among patients who receive autogenous vein grafts to treat chronic critical limb ischemia; on the occurrence of clinically significant graft stenosis (more than or equal to 70%); and on the incidence of critical limb ischemia (e.g., gangrene, non-healing ischemic ulcers or ischemic rest pain).

DETAILED DESCRIPTION:
Peripheral vascular disease manifested by narrowing of the peripheral arteries is one of the more common manifestations of atherosclerotic vascular disease. Complications such as claudication, rest pain, and impaired wound healing are frequent and may result in gangrene and amputation. Restoration of circulation to the lower extremities may be undertaken using a variety of techniques including angioplasty, stenting, and bypass grafting.

Approximately 99,000 infra-inguinal bypass procedures were performed in the U.S. in 1998. It is estimated that approximately 22% of all infra-inguinal bypass grafts will fail by 12 months. Graft failure rates have been estimated to increase to 40% at 12 months for patients receiving composite, cephalic or lesser saphenous (high-risk) vein grafts (Vascular Surgery Registry, Brigham and Women's Hospital). These primary graft failures are typically due to stenoses that result from neointimal hyperplasia, a pathological adaptation process that occurs in veins exposed to the arterial circulation. The consequences of graft failure are as significant as those of primary atherosclerotic disease and include ischemia and poor wound healing that may result in amputation. Since the long-term patency of venous grafts can be improved with treatment prior to frank occlusion, considerable efforts have been focused on the methods for the detection of grafts at high-risk for failure. Duplex ultrasonography has been determined to be a sensitive screening test for the early detection of failing grafts. Peak systolic velocity (PSV), as measured by duplex ultrasound, has been shown to be a sensitive marker for low flow, and wave form analysis has permitted the identification of areas of stenosis in the vein under study. Management of patients who have undergone infra-inguinal bypass therefore includes routine surveillance with duplex ultrasound and the immediate correction of significant (more than or equal to 70%) graft stenoses.

ELIGIBILITY:
PATIENTS MUST:

* Be scheduled to undergo infra-inguinal bypass grafting surgery using excised autogenous vein for Chronic Critical Limb Ischemia (i.e., rest pain, non-healing ulceration or gangrene). For patients presenting with rest pain as the only manifestation of CCLI, must have the diagnosis confirmed by at least one of the following,: i.) an ankle pressure of < 50 mmHg (or ABI <0.4), ii.) a toe pressure < 30 mmHg, iii.) a reduced TCPO2 < 30 mmHg, or iv.) a severely ischemic or flat line transtarsal pulse volume recording (i.e., Category V).
* Be males or females of at least 18 years old.
* Have agreed to participate voluntarily and signed and dated an IRB-approved, Patient Informed Consent form.
* Have a documented negative serum pregnancy test for all women of childbearing potential.
* Be using an acceptable method of birth control if of reproductive potential.
* Note: Patients undergoing operations to replace previously occluded grafts that involve placement of an entirely new bypass graft ARE eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400
Dates: Start 2001-11; Study Completion 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Todd Lorenz, M.D., Study Director — Anesiva, Inc.
Locations (121):
- United States (114):
  - The Kirklin Clinic, Birmingham, Alabama
  - University Hospital, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Vascular Specialists of Mobile, PC, Mobile, Alabama
  - Springhill Memorial Hopsital, Mobile, Alabama
  - Tucson Heart Hospital, Tucson, Arizona
  - University Medical Center, Tucson, Arizona
  - Northwest Hospital, Tucson, Arizona
  - Tucson Vascular Surgery, Tucson, Arizona
  - Southern Arizona Vascular Institute, Tucson, Arizona
  - St. Mary's Hospital, Tucson, Arizona
  - Baptist Health, Little Rock, Arkansas
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences Hospital, Little Rock, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - San Diego, SCPMG, Department of Surgery, San Diego, California
  - Kaiser Permanente Franklin Medical Center, Denver, Colorado
  - Exempla Healthcare Saint Joseph Hospital, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Washington Hospital Center, Center for Vascular Care, Washington D.C., District of Columbia
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Samson Showalter Vascular Specialists, Sarasota, Florida
  - Clinical Research Center, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Vascular & Surgery Assoc., Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University School of Medicine Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Vascular Institute of Georgia, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Methodist Hospital, Indianapolis, Indiana
  - Veteran's Affairs Medical Center, Indianapolis, Indiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dept. of Surgery at Harvard Medical Faculty Physicians, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - O.W. Brown, M.D., Southfield, Michigan
  - Steven D. Rimar, M.D., Troy, Michigan
  - St. Mary's Hospital, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Methodist Hospital, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dr. Randy Shafrtiz, Clinical Office, Holmdel, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Surgical Specialists of NJ, Morris Vascular Center, Morristown, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Umdnj-Rwjms, New Brunswick, New Jersey
  - UMDNJ - New Jersey Medical School, University Hospital, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Kings County Hospital, Brooklyn, New York
  - SUNY Downstate University Hospital of Brooklyn and Medical School, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - New York Presbyterian Hospital, Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Hospital, The Bronx, New York
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Department of Surgery, Division of Vascular Surgery, East Carolina University, Greenville, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Jobst Vascular Center, Toledo, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Veterans Administration Healthcare System, Pittsburgh, Pennsylvania
  - Robert Packer Hospital, Sayre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina Hospital, Charleston, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - St. Thomas Medical, Nashville, Tennessee
  - The Surgical Group, PLLC, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - VAMC, Houston, Texas
  - University Medical Center, Lubbock, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Baptist Medical Center, San Antonio, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - Northeast Baptist Hospital, San Antonio, Texas
  - Pro-Research Group, San Antonio, Texas
  - Southwest Texas Methodist Hospital, San Antonio, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Vascular and Transplant Specialists, Peripheral Vascular Laboratory, Chesapeake, Virginia
  - Vascular and Transplant Specialsts, Peripheral and Vascular Laboratory, Chesapeake, Virginia
  - Southampton Memorial Hospital, Franklin, Virginia
  - Shore Memorial Hospital, Nassawadox, Virginia
  - Chesapeake General Hospital, Norfolk, Virginia
  - Vascular and Transplant Specialists, Peripheral Vascular Laboratory, Norfolk, Virginia
  - Virginia Vascular Associates, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Jefferson Surgical Clinic, Roanoke, Virginia
  - Harborview Medical Center, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Froedert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Clement J. Zablocki VAMC, Milwaukee, Wisconsin
- Canada (7):
  - Peter Lougheed Centre, Calgary, Alberta
  - Vancouver Hospital & Health Sciences Centre, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - St. Paul's Hospital, Saskatoon, Saskatchewan